CLINICAL TRIAL: NCT04807400
Title: A Phase IIIb, Multicentre, Randomised Controlled Study to Evaluate the Implementation, Preference and Utility for Administration of Inclisiran Sodium in Participants With Atherosclerotic Cardiovascular Disease (ASCVD) or ASCVD-risk Equivalents and Elevated Low Density Lipoprotein Cholesterol (LDL-C) Using a Primary Care Models in the NHS.
Brief Title: Study in Primary Care Evaluating Inclisiran Delivery Implementation + Enhanced Support
Acronym: SPIRIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CKJX839A1GB01; 2020-004401-31 (EudraCT Number)
Record Dates: First submitted 2021-03-17; First posted 2021-03-19 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Atherosclerotic Cardiovascular Disease; Atherosclerotic Cardiovascular Disease Risk Equivelents; Elevated Low Density Lipoprotein Cholesterol
Keywords: Atherosclerotic Cardiovascular Disease; Atherosclerotic Cardiovascular Disease Risk Equivalents; Elevated Low Density Lipoprotein Cholesterol; ASCVD; LDL-C
MeSH Terms: conditions — Atherosclerosis | interventions — ALN-PCS

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control+ BS (Active Comparator): Participants continued to receive their background lipid lowering therapy plus behavioural support (BS).
  Interventions: Behavioral: Behavioural Support; Drug: Background lipid lowering therapy
- Inclisiran (Experimental): Participants continue to receive their background lipid lowering therapy, plus inclisiran for injection (delivered in an injection-only model).
  Interventions: Drug: Inclisiran; Drug: Background lipid lowering therapy
- Inclisiran + BS (Experimental): Participants continued to receive their background lipid lowering therapy, plus inclisiran for injection, plus behavioural support.
  Interventions: Drug: Inclisiran; Behavioral: Behavioural Support; Drug: Background lipid lowering therapy

INTERVENTIONS:
Drug: Inclisiran — Inclisiran Sodium 300mg on Day 1 and Day 90 by subcutaneous injection
  Arms: Inclisiran; Inclisiran + BS
Behavioral: Behavioural Support — Regular telephone based behavioural support programme delivered throughout the study period, as measured by point of care testing device.
  Arms: Control+ BS; Inclisiran + BS
Drug: Background lipid lowering therapy — lipid-lowering therapy (such as a statin and/or ezetimibe) as background therapy

SUMMARY:
The purpose of this study was to evaluate the implementation of inclisiran in a regional primary care setting in the UK

Inclisiran, also known as KJX839, is a medication made to reduce the level of "bad" cholesterol (LDL-cholesterol) in the blood. Inclisiran works in a way that makes the liver produce less of a substance called 'PCSK9'. PCSK9 reduces the ability of the liver to remove LDL-cholesterol from the blood. By lowering the production of PCSK9, Inclisiran leads to more LDL-cholesterol being removed by the liver from the blood, thereby reducing LDL-cholesterol overall.

DETAILED DESCRIPTION:
A phase IIIb, multicenter, randomized controlled study to evaluate the implementation, preference, and utility for administration of inclisiran sodium in participants on established lipid lowering medication or, have been recommended lipid lowering therapy by their healthcare provider but are unable to tolerate treatment, with elevated low density lipoprotein cholesterol (LDL-C) in a primary care population. This study was an implementation research study that utilized implementation science methodology and use of the electronic medical record (EMR).

Using implementation science methodology, the study intended to assess the effect of 9 months treatment with inclisiran with/without behavioural support, compared to standard of care + behavioural support, on LDL-C reduction, total lipid profile, assessments of patient and healthcare professional (HCP) satisfaction, health-care resource utilization and healthcare service process evaluation.

The primary focus of this study was implementation and 'transactability' - how to organize, deliver and maintain an innovative treatment for Atherosclerotic Cardiovascular Disease (ASCVD) in a primary care setting in a sustainable way.

Patients taking part in the study were randomised to one of three groups:

* Control + BS: Participants continued to receive their background lipid lowering therapy plus behavioural support. Subjects in treatment group 1 were referred to as the control group in this study
* Inclisiran: Participants continue to receive their background lipid lowering therapy, plus inclisiran for injection (delivered in an injection-only model).
* Inclisiran + BS: Participants continued to receive their background lipid lowering therapy, plus inclisiran for injection, plus behavioural support.

Participants who were randomized to Inclisiran or Inclisiran + BS received one injection of inclisiran on Day 1 and a second injection of inclisiran on Day 90.

Participants in Control + BS and Inclisiran + BS received a monthly telephone call from a health advisor, providing support to enable participants to make positive behaviour changes to reduce their cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent had to be obtained prior to participation in the study.
2. Patients on established lipid lowering medication or, have been recommended lipid lowering therapy by their health care provider but were unable to tolerate treatment.
3. A total cholesterol measurement at screening that was ≥4 mmol/L [approximately 160 mg/dL].
4. Participants on lipid-lowering therapies had to be on a stable dose for ≥30 days before screening with no planned medication or dose change.

Exclusion Criteria:

1. Medical or surgical history that might limit the individual's ability to take study treatments for the duration of the study and/or put the participant at significant risk .
2. Current or planned renal dialysis or transplantation.
3. Acute coronary syndrome or stroke less than 4 weeks before the screening visit.
4. Coronary revascularization procedure planned within the next 6 months.
5. Women of child-bearing potential, unless they agree to abstinence or, if sexually active, agree to the use of effective methods of contraception during the study.
6. Women who are pregnant or breast-feeding.
7. Previous, current or planned treatment with a monoclonal antibody targeting PCSK9, or with a drug known to be contra-indicated with inclisiran.
8. Previous exposure to inclisiran or participation in a randomised study of inclisiran.
9. Current or previous participation in a clinical study with an unlicensed drug or device within 30 days or five half-lives of the screening visit, whichever is longer.
10. Participants who planed to move away from the geographical area where the study is being conducted during the study period.
11. A triglyceride measurement at screening that is greater than or equal to 4.52 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United Kingdom (13):
  - Novartis Investigative Site, Sale, Cheshire
  - Novartis Investigative Site, Altrincham, Manchester
  - Novartis Investigative Site, Davyhulme, Manchester
  - Novartis Investigative Site, Didsbury, Manchester
  - Novartis Investigative Site, Northenden, Manchester
  - Novartis Investigative Site, Sale, Manchester
  - Novartis Investigative Site, Swinton, Manchester
  - Novartis Investigative Site, Wythenshawe, Manchester
  - Novartis Investigative Site, Chadderton
  - Novartis Investigative Site, Cheadle Hulme
  - Novartis Investigative Site, Greater Manchester
  - Novartis Investigative Site, Lancashire
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wilson P, Elvey R, Mathieson A, Bower P, Gibson M, Vell T, Dixon S. Evaluating the implementation of inclisiran in primary care: process evaluation interim findings from interviews with key stakeholders. BMJ Open. 2025 Feb 26;15(2):e083441. doi: 10.1136/bmjopen-2023-083441. PMID 40010816
- [Derived] Mathieson A, Elvey R, Wilson P. Development and application of a qualitative rapid analysis framework in a hybrid trial within primary care. BMJ Open. 2024 Jul 24;14(7):e076792. doi: 10.1136/bmjopen-2023-076792. PMID 39053958
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2082

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 17 primary care centres with a network of research ready General Practitioners across Greater Manchester, United Kingdom.
Pre-assignment Details: Eligibility and recruitment to the study was optimized by using NorthWest EHealth's (NWEH) proven Feasibility Assessment and Recruitment System for Improving Trial Efficiency (FARSITE) for identification and recruitment at participating General Practitioner practices.
Period: Overall Study
Arm/Group | Inclisiran | Inclisiran + BS | Control+ BS
Started | 298 | 297 | 297
Full Analysis Set (Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug.) | 297 (There was one patient who was mistakenly randomized despite not meeting the predefined exclusion criteria; however, this patient did not receive the study treatment and was excluded from the full analysis set as per the definition.) | 297 | 297
Safety Set (Safety Set comprised all participants who received at least one dose of study treatment.) | 273 | 281 | 290
Completed | 248 | 252 | 234
Not Completed | 50 | 45 | 63
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Death | 2 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 6
Not completed — Non-Compliance With Study Drug | 0 | 4 | 1
Not completed — Participant Decision | 20 | 19 | 26
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 4 | 3 | 7
Not completed — Withdrawal by Subject | 13 | 9 | 20
Not completed — Mis-randomized | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Participants are based on the Full Analysis Set (FAS) population, as primary and secondary analysis are based on the FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | Inclisiran | Inclisiran + BS | Control+ BS | Total
Number analyzed (Participants) | 297 | 297 | 297 | 891
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.0 (9.27) | 65.8 (9.71) | 66.7 (9.45) | 66.2 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 174 | 180 | 524
  Male | 127 | 123 | 117 | 367
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 11 | 3 | 9 | 23
  Black | 1 | 0 | 5 | 6
  Mixed | 1 | 3 | 1 | 5
  White | 281 | 289 | 278 | 848
  Other | 3 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline to Day 270
Description: Change in Low Density Lipoprotein Cholesterol (LDL-C) after 270 days of treatment in adults on established lipid lowering medication or who have been recommended lipid lowering therapy by their health care provider but are unable to tolerate treatment, regardless of treatment discontinuation for any reason and regardless of unforeseen change in the concomitant lipid lowering therapy.
  Multiple imputation is used to impute missing data using a washout model.
Time Frame: Baseline, Day 270
Population: Full analysis set. The Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug. Only participants with LDL-C values at both, baseline and Day 270, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline in LDL-C
Arm/Group | Inclisiran | Inclisiran + BS | Control+ BS
Number analyzed (Participants) | 294 | 295 | 293
percent change from baseline in LDL-C | -37.3 (2.29) | -37.6 (2.33) | -5.4 (2.34)
Statistical Analysis 1: Comparison: Inclisiran vs Control+ BS; Test type: Superiority; p < 0.001, ANCOVA — p-values are adjusted using Holm's procedure; Least Squares Mean = -31.8, 95% CI 2-sided [-37.91 to -25.77], Standard Error of Mean 3.10
Statistical Analysis 2: Comparison: Inclisiran + BS vs Control+ BS; Test type: Superiority; p < 0.001, ANCOVA — p-values are adjusted using Holm's procedure; Least Squares Mean = -32.1, 95% CI 2-sided [-38.35 to -25.94], Standard Error of Mean 3.17

2. Secondary Outcome: Number of Participants Interviewed for CFIR Analysis.
Description: To identify the need to support the implementation of inclisiran in the real world, a framework was drawn known as the Consolidated Framework for Implementation Research (CFIR). Patients who received inclisiran were interviewed to understand their experience with the program and to obtain a comprehensive understanding, with or without behavioural support. These patients were interviewed on various aspects of their experience related to their high cholesterol management, trial participation, inclisiran injections, attending appointments, and if applicable their experience with the behavioural support programme.
  These interviews were not set up in a way that allow numerical analysis. The process evaluation was conducted by Manchester University.
Time Frame: Day 270
Population: All patients randomized to inclisiran
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran | Inclisiran + BS
Number analyzed (Participants) | 297 | 297
Participants | 28 | 28

3. Secondary Outcome: Patient Reported Outcomes: CSQ-8 Total Score After Treatment
Description: The Client Satisfaction Questionnaire (CSQ)-8 is the standard self-administered CSQ scale containing 8 items that comprise the measurement of satisfaction with services and measurement of improvement of capacity to cope and change adaptively. Items include questions enquiring about respondents' opinions and conclusions about services they have received or are currently receiving. Response options differ from item to item, but all are based on a four-point scale. For the CSQ-8 version, scores range from 8 to 32, with higher values indicating higher satisfaction.
Time Frame: Day 90
Population: Full analysis set: The Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug. Only participants with CSQ-8 assessment Day 90, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Inclisiran | Inclisiran + BS | Control+ BS
Number analyzed (Participants) | 160 | 163 | 105
score on a scale | 30.1 (0.24) | 30.1 (0.24) | 28.7 (0.30)
Statistical Analysis 1: Comparison: Inclisiran vs Control+ BS; Test type: Superiority; p < 0.001, ANOVA; Least-squares Mean = 1.4, 95% CI 2-sided [0.62 to 2.13], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Inclisiran + BS vs Control+ BS; Test type: Superiority; p < 0.001, ANOVA; Least-squares Mean = 1.3, 95% CI 2-sided [0.60 to 2.10], Standard Error of Mean 0.38

4. Secondary Outcome: Patient Reported Outcomes: CSQ-8 Total Score Between Inclisiran Arms
Description: The CSQ-8 is the standard self-administered CSQ scale containing 8 items that comprise the measurement of satisfaction with services and measurement of improvement of capacity to cope and change adaptively. Items include questions enquiring about respondents' opinions and conclusions about services they have received or are currently receiving. Response options differ from item to item, but all are based on a four-point scale. For the CSQ-8 version, scores range from 8 to 32, with higher values indicating higher satisfaction.
  This secondary outcome only analysed data of the two Inclisiran arms, by considering the Inclisiran only arm as the control group. The standard error for Least Square Mean could change because dropping a treatment arm affects the estimation of treatment effects and the variability of data.
Time Frame: Day 90
Population: Full analysis set: The Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug. Only participants assigned to inclisiran with CSQ-8 assessment Day 90, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Inclisiran + BS | Inclisiran
Number analyzed (Participants) | 163 | 160
score on a scale | 30.1 (0.23) | 30.1 (0.23)
Statistical Analysis 1: Comparison: Inclisiran + BS vs Inclisiran; Test type: Superiority; p = 0.9347, ANOVA; Least-squares Mean = -0.03, 95% CI 2-sided [-0.67 to 0.61], Standard Error of Mean 0.326

5. Secondary Outcome: Change From Baseline to Day 90 in Total PAM Score
Description: The Patient Activation Measure (PAM) questionnaire is a survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare.
  This study used the 13-point PAM questionnaire, which consists of 13 statements relating to patients beliefs about health care, confidence in their management of health related tasks, and self-assessed knowledge of their condition. For each statement patients are required to say how much they either agree or disagree on a response scale of 1-5, where 1 represents "strongly disagree", 4 represents "strongly agree" and 5 indicates that the statement is "not applicable" to them. A standardised spreadsheet in excel is used to score the PAM. Responses are used to generate a continuous score from 0 to 100 where higher scores indicate that the patient is more activated.
Time Frame: Baseline, Day 90
Population: Full analysis set: The Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug. Only participants with PAM assessment at both, Baseline and Day 90, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Inclisiran | Inclisiran + BS | Control+ BS
Number analyzed (Participants) | 108 | 115 | 37
score on a scale | 2.4 (1.18) | 2.7 (1.14) | 1.4 (2.01)
Statistical Analysis 1: Comparison: Inclisiran vs Control+ BS; Test type: Superiority; p = 0.6759, ANCOVA; Least-squares Mean = 1.0, 95% CI 2-sided [-3.62 to 5.58], Standard Error of Mean 2.34
Statistical Analysis 2: Comparison: Inclisiran + BS vs Control+ BS; Test type: Superiority; p = 0.5756, ANCOVA; Least-squares Mean = 1.3, 95% CI 2-sided [-3.25 to 5.84], Standard Error of Mean 2.31

6. Secondary Outcome: Change From Baseline to Day 90 in Total PAM Score Between Inclisiran Arms
Description: The Patient Activation Measure (PAM) questionnaire is a survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare. This study used the 13-point PAM questionnaire, which consists of 13 statements. For each statement patients are required to say how much they either agree or disagree on a response scale of 1-5, where 1 represents "strongly disagree", 4 represents "strongly agree" and 5 indicates that the statement is "not applicable" to them. Responses are used to generate a continuous score from 0 to 100 where higher scores indicate that the patient is more activated.
  This outcome only analysed data of the two inclisiran arms, by considering the Inclisiran only arm as the control group. In an ANCOVA model, the Least Squares Means and corresponding Standard Error could change because the removal of a treatment group affects the estimation of the treatment effects and the adjustment for the covariate(s).
Time Frame: Baseline, Day 90
Population: Full analysis set: The Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug. Only participants assigned to inlcisiran with PAM assessment at Day 90, were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Inclisiran + BS | Inclisiran
Number analyzed (Participants) | 115 | 108
score on a scale | 2.6 (1.17) | 2.3 (1.21)
Statistical Analysis 1: Comparison: Inclisiran + BS vs Inclisiran; Test type: Superiority; p = 0.8580, ANCOVA; Least-squares Mean = 0.3, 95% CI 2-sided [-3.02 to 3.62], Standard Error of Mean 1.69

7. Secondary Outcome: Measures of Adherence to Cardiovascular Disease Self-management Using the Validated Patient Activation Measure (PAM) Questionnaire.
Description: The Patient Activation Measure (PAM) questionnaire is a survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or her own health and healthcare.
  This study used the 13-point PAM questionnaire, which consists of 13 statements relating to patients beliefs about health care, confidence in their management of health related tasks, and self-assessed knowledge of their condition. For each statement patients are required to say how much they either agree or disagree on a response scale of 1-5, where 1 represents "strongly disagree", 4 represents "strongly agree" and 5 indicates that the statement is "not applicable" to them. Responses are used to generate a continuous score from 0 to 100.
  The continuous PAM scores are then categorised into 4 levels: Level 1 - disengaged and overwhelmed; Level 2 - become aware but still struggling; Level 3 - taking action; Level 4 - maintaining behaviors and pushing further.
Time Frame: Baseline, Day 90
Population: Full analysis set: The Full Analysis Set (FAS) comprised of all randomized participants except for those mis-randomized participants who did not receive study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Inclisiran | Inclisiran + BS | Control+ BS
Number analyzed (Participants) | 297 | 297 | 297
Participants
  Level 1 (Disengaged and overwhelmed) at Baseline | 13 | 20 | 7
  Level 2 (Become aware but still struggling) at Baseline | 47 | 50 | 15
  Level 3 (Taking action) at Baseline | 61 | 75 | 36
  Level 4 (Maintaining behaviors and pushing further) at Baseline | 48 | 44 | 21
  Missing PAM scores at baseline | 128 | 108 | 218
  Level 1 (Disengaged and overwhelmed) at Day 90 | 9 | 8 | 6
  Level 2 (Become aware but still struggling) Day 90 | 37 | 38 | 23
  Level 3 (Taking action) at Day 90 | 63 | 64 | 46
  Level 4 (Maintaining behaviors and pushing further) at Day 90 | 56 | 47 | 33
  Missing PAM scores at Day 90 | 132 | 140 | 189

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study visit plus 30 days post treatment, up to a maximum duration of 300 days.
Description: Any sign or symptom that occurs during the conduct of the trial and the safety follow-up.
Groups:
- Control + BS: Participants continued to receive their background lipid lowering therapy plus behavioural support (BS).
- Total: Total
Arm/Group | Inclisiran | Inclisiran + BS | Control + BS | Total
All-Cause Mortality (participants affected / at risk) | 2/273 | 0/281 | 0/290 | 2/844
Serious Adverse Events (participants affected / at risk) | 24/273 | 36/281 | 28/290 | 88/844
Other Adverse Events (participants affected / at risk) | 3/273 | 2/281 | 0/290 | 5/844
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=273) | Inclisiran + BS (N=281) | Control + BS (N=290) | Total (N=844)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 2 | 4
Angina unstable (Cardiac disorders) | 1 | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 5 | 0 | 7
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 2
Left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Acquired oesophageal web (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Chest pain (General disorders) | 0 | 1 | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Biliary sepsis (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2 | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 2
Localised infection (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 4 | 1 | 1 | 6
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 3
Urosepsis (Infections and infestations) | 1 | 2 | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 1 | 0 | 1
Platelet count abnormal (Investigations) | 0 | 0 | 1 | 1
White blood cell count abnormal (Investigations) | 0 | 0 | 1 | 1
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1 | 2 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Chronic lymphocytic leukaemia stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Bell's palsy (Nervous system disorders) | 1 | 0 | 0 | 1
Carotid artery dissection (Nervous system disorders) | 0 | 1 | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Psychotic symptom (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 0 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal mass (Renal and urinary disorders) | 0 | 1 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 1 | 1 | 2
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inclisiran (N=273) | Inclisiran + BS (N=281) | Control + BS (N=290) | Total (N=844)
Injection site rash (General disorders) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04807400/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04807400/SAP_001.pdf